CLINICAL TRIAL: NCT07400926
Title: Clinical In-use Observational Trial to Evaluate the Updated Inserter for the Travoprost Intracameral Implant 75 mcg
Brief Title: Observational Trial of the Updated Inserter for the Travoprost Intracameral Implant 75mcg
Acronym: TRIO
Status: Recruiting | Type: Observational
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GLK-101-03
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Open-angle Glaucoma, Ocular Hypertension
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Travoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Model G2-TRIO: Subjects receive a Travoprost intracameral implant with the Model G2-TRIO
  Interventions: Combination Product: Travoprost

INTERVENTIONS:
Combination Product: Travoprost — Travoprost intracameral implant, 75mcg administered using the sterile, single-dose updated inserter (Model G2-TRIO)

SUMMARY:
Clinical in-use observational trial to evaluate the updated inserter for the Travoprost Intracameral implant using the updated inserter (Model G2-TRIO)

DETAILED DESCRIPTION:
The objective of this study is to evaluate the administration of the Travoprost intracameral implant using the updated inserter (Model G2-TRIO)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Open-angle glaucoma
* 18 years of age or older

Exclusion Criteria:

* Subject who is breast-feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with OAG or OHT
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Successful implantation | 1 day
  Investigator's ability to follow the Instructions For Use/Prescribing Information and correctly administer the model G2-TRIO travoprost intracameral implant 75mcg with the updated inserter

CONTACTS AND LOCATIONS:
Locations (1):
- Glaukos Investigative Site, Kenosha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No